CLINICAL TRIAL: NCT03698981
Title: Randomized Controlled Trial to Reduce Stigma and Improve Treatment Adherence in HIV+ Pregnant Women in Botswana
Brief Title: Reduce Stigma and Improve Treatment Adherence in HIV+ Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TW011084-01
Record Dates: First submitted 2018-09-05; First posted 2018-10-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: HIV; Stigma
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: To account for expected drop out (~10%), ~220 participants will be recruited, resulting in MME and TAU groups of ~100 with complete data by the 56th week following the beginning of pregnancy. For the MME arm, we will enroll 9-10 women per group on a rolling basis to comprise ~12 intervention groups total; ~1 MME group will be initiated per month.
Who Masked: Outcomes Assessor
Masking Description: Staff conducting "primary outcome measures" with mothers at baseline, post-intervention, and week 56 (in person) will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers Moving towards Empowerment (MME) (Experimental): The MME intervention arm will complete our 8-session intervention, weekly for 60-70 minutes per session. Homework will be assigned each week and reviewed the next session. Certificates will be issued to participants who complete the intervention. Fidelity assessments for each session will be evaluated by local research personnel.
  Interventions: Behavioral: Mothers Moving towards Empowerment (MME)
- Treatment As Usual (TAU) (No Intervention): Control condition participants will receive Treatment as usual (TAU), including using free ART and antenatal services as they wish. Control condition participants are assessed on all 'Primary outcomes' at the same time points as the MME intervention group.

INTERVENTIONS:
Behavioral: Mothers Moving towards Empowerment (MME) — MME integrates 3 components: 1) psychoeducation regarding causes, transmission, and treatment of HIV re how adherence to ART and antenatal care acts to promote health for HIV+ women and PMTCT82,83. We will emphasize ART adherence spanning into PP as a maternal duty to raise a healthy child; 2) challenging stereotypes of HIV+ women, such as promiscuity, that threaten core aspects of being a "good woman" and hinder treatment adherence; 3) coping skills for HIV-related discrimination, i.e., rejection or abandonment by male partners leading to discontinuing treatment adherence and impacts on raising children.
  Arms: Mothers Moving towards Empowerment (MME)

SUMMARY:
The goal of this proposal is to use a theoretically grounded approach to culturally-tailor a stigma intervention among just identified, pregnant HIV+ women in Botswana. This project will use empirically tested stigma interventions that have shown efficacy for serious mental illness and to adapt these to HIV. Additionally, a novel component of this intervention is the utilization of peers (i.e., mothers with HIV), which has been shown to be an effective stigma reduction agent for other conditions but has not yet been widely used with HIV.

The investigators propose to leverage this middle-income context to conduct a Randomized Controlled Trial (RCT) with HIV+ women (n=100 intervention group, n=100 control group). The investigators examine the stigma intervention for outcomes among mothers (including adherence to Antiretroviral therapy [ART] and antenatal treatment), and conduct exploratory birth outcomes among infants (e.g., birth weight, time of delivery) as well. Capacity building activities to transfer stigma intervention knowledge will occur throughout the project to enable investigators in Botswana to independently develop stigma interventions, thus serving as a model for other African countries. Finally, this pilot intervention will provide valuable data for future intervention trials to reduce stigma and improve ART adherence.

DETAILED DESCRIPTION:
To be completed by University of Botswana Research team:

The investigators will sample from the Dept. of Obstetrics and Gynecology (OB/GYN) at Princess Marina Hospital IDCC. Newly-diagnosed pregnant HIV+ women are referred to OB care at Ministry of Health (MOH) antenatal clinics and receive HIV care at the IDCC for continued ART. To account for expected drop out (~10%), ~220 participants will be recruited. All participants will be randomized to receive MME (the HIV-stigma intervention) or TAU (treatment as usual) from week 28-36 of their pregnancy. The investigators will initiate MME in the antenatal period because the cultural practice of botsetsi (below) could impede implementation post-partum. All participants will have PMTCT by initiation of ART before week 32. Adherence to ART, antenatal and PP care, and viral load testing will be tracked from week 28 of pregnancy to 16 weeks PP (~week 56 for full-term babies).

Procedures. To account for expected drop out (~10%), ~220 participants will be recruited, resulting in MME and TAU groups of ~100 with complete data at week 56. For the MME (intervention) arm, the investigators will enroll 9-10 women per group on a rolling basis to comprise ~12 intervention groups total; ~1 MME group will be initiated per month.

Intervention & Assessment Procedures. One advantage of our study is that, whenever possible, the investigators augment self-report measures with objective measures from medical records (i.e., for infants, birth-weights, APGAR scores at birth; for antenatal treatment, an Antenatal/delivery record tracking antenatal visits that is filled out by doctors; for ART, CD4 count and Viral load data from the integrated patient management system). Fidelity assessments for each session will be evaluated by Ho-Foster. Control Description: Control condition participants will receive TAU, including using free ART and antenatal services as they wish. Control condition participants are assessed on all 'Primary outcomes' at the same time points as the intervention group.

Follow-up Assessment (Months 18-22): Mothers' Postpartum (PP) adherence (56 weeks) serves as a key outcome. The investigators examine a set of exploratory, infant birth outcomes that may result from improved antenatal care and ART adherence. The investigators use an "Under 5 (years old) card" that is filled out by a doctor to track infant's developmental outcomes which is carried by the mother. Child outcomes include: APGAR score, preterm delivery, mortality (at <16 weeks), birthweight, vaccination record, and mother-to-child-transmission of HIV (MTCT). The investigators will call each participant at 4 months' time and ask to meet in person to review their "Under 5 card" to record infant outcomes at both: a) time of birth; b) 16 weeks PP.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women
* aged 18 to 45
* diagnosed as HIV+
* receiving care through IDCC with Botswana citizenship
* speak either English or Setswana
* able to provide informed consent

Exclusion Criteria:

* unable to provide informed consent
* non-English or Setswana speakers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All participants must be Primiparous women diagnosed as HIV+ receiving both antenatal care and ART.
Enrollment: 59 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Internalized Stigma | 7 minutes
  Assesses extent HIV stereotypes are applied to the self. 18 items. (scale 0-3). Good reliability & validity
Anticipated Stigma | 4 minutes
  Assesses extent people living with HIV/AIDS (PLWHA) anticipate rejection if HIV disclosed. 10 items. (scale 0-3) Good reliability & validity
Perceived Community Stigma | 8 minutes
  Assesses extent community members would devalue PLWHA. 20 items (scale: 0-3) Good reliability & validity
Enacted Stigma | 10 minutes
  Experienced stigma by PWLHA. 28 items. (scale 0-3). Good reliability & validity

SECONDARY OUTCOMES:
APGAR Score | 1minute
  Objective: 0-10 as rated by physician (documented at 5 minutes and 10 minutes)
Pre-term delivery | 1minute
  Objective: Born prior to 37 weeks or 37 weeks and after (Yes/ No). Check hospital record
Mortality | 1minute
  Objective: Mortality (e.g. neonatal, infant mortality) (Yes/No). Check hospital record
Birthweight | 1minute
  Objective: Infant weight in grams (low = <2500 g or normal = >2500 g)
Vaccinations | 1minute
  Objective: from 0-4 visits; Vaccines given at 0, 2, 3, and 4 months (e.g., BCG's, Hep B) (score: 0-3 months)
Infant HIV status | 1minute
  PCR Assay conducted at 6 weeks and reflected in medical record; (Y/N)

OTHER OUTCOMES:
Quality of Life Assessment scale | 16 minutes
  Self-report scale assessing quality of life. 42 items (scale 0-4). Good reliability & validity.
Depressive Sx-CES-D | 8 minutes
  Self-report scale assessing depressive symptoms. 20 items (scale 0-3). Good reliability & validity
Social Support | 16 minutes
  Self-report scale assessing functional social support. 40 items (scale 0-3). Good reliability & validity

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Yang, Ph.D., Principal Investigator — New York University
Locations (1):
- Princess Marina Hospital IDCC, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Poku OB, Ho-Foster AR, Entaile P, Misra S, Mehta H, Rampa S, Goodman M, Arscott-Mills T, Eschliman E, Jackson V, Melese T, Becker TD, Eisenberg M, Link B, Go V, Opondo PR, Blank MB, Yang LH. 'Mothers moving towards empowerment' intervention to reduce stigma and improve treatment adherence in pregnant women living with HIV in Botswana: study protocol for a pragmatic clinical trial. Trials. 2020 Oct 7;21(1):832. doi: 10.1186/s13063-020-04676-6. PMID 33028387